CLINICAL TRIAL: NCT05655611
Title: Effects Of Muscle Energy Technique With Or Without First Rib Mobilization On Range Of Motion And Pain In Adhesive Capsulitis
Brief Title: Muscle Energy Technique With Or Without First Rib Mobilization In Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AH/21/0130/SIDRA
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Adhesive Capsulitis
Keywords: muscle energy technique, first rib mobilization
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- first rib mobilization (Experimental): To perform the first rib mobilization, the patient remained lying supine with the head in the examiner's right hand. Examiner then palpated the left first rib and passively side-bended the patient's head to the left to relieve any muscular tension on the first rib. Patient was then asked to take a deep breath in and out. During exhalation, the examiner applied pressure to depress the first rib, holding it in place at the end of the exhalation. Then, holding the first rib in place, the patient was asked to inhale and exhale deeply again. The examiner continued applying pressure to hold the first rib in a position of relative depression during inhalation, and further depressed the first rib as able during exhalation. This process was repeated three times in two sets, for a total of six first rib depression mobilizations
  Interventions: Other: first rib mobilization
- muscle energy technique (Active Comparator): All the patients will receive conventional physical therapy treatment and muscle energy techniques for shoulder flexion, abduction, internal and external rotation. Muscle energy technique was applied for five repetitions per set, five sets per session, one session per day, three days a week for three weeks with each repetition maintained for the duration of 7-10 seconds
  Interventions: Other: muscle energy technique

INTERVENTIONS:
Other: first rib mobilization — To perform the first rib mobilization, the patient remained lying supine with the head in the examiner's right hand. Examiner then palpated the left first rib and passively side-bended the patient's head to the left to relieve any muscular tension on the first rib. Patient was then asked to take a deep breath in and out. During exhalation, the examiner applied pressure to depress the first rib, holding it in place at the end of the exhalation. Then, holding the first rib in place, the patient was asked to inhale and exhale deeply again. The examiner continued applying pressure to hold the first rib in a position of relative depression during inhalation, and further depressed the first rib as able during exhalation. This process was repeated three times in two sets, for a total of six first rib depression mobilizations.
  Other Names: first rib maitland mobilization
  Arms: first rib mobilization
Other: muscle energy technique — Muscle energy technique for glenohumeral joint restricted abduction-The therapist stood in front of the patient, then placed one hand over the top of the subject's involved shoulder. The therapist cups the glenohumeral joint to palpate for motion and the subjects are directed to press the elbow towards their body. Muscle energy technique was applied for five repetitions per set, five sets per session, one session per day, three days a week for three weeks with each repetition maintained for the duration of 7-1 seconds.
  Other Names: muscle energy technique for shoulder
  Arms: muscle energy technique

SUMMARY:
This study will be a randomized control trial. Study will be conducted in 40 patients in the age range 40-70 years, which will be selected by using non proability convenient sampling technique. Subjects will be divided in 2 groups. Group A will receive first rib mobilization along with METS and conventional treatment, group B will receive METS and conventional physical therapy treatment only. Treatment will be given thrice per week for 3 weeks. Data will be collected pre and post treatment, for data collection numeric pain rating scale, shoulder pain and disability index (SPADI) will be used. Joint range of motion will be measured using goniometer. After collection data from defined study setting, data will be entered and analyzed at Riphah International University, Lahore.

DETAILED DESCRIPTION:
Adhesive capsulitis, also known as "frozen shoulder," is a common condition of the shoulder defined as a pathologic process in which contracture of the gleno-humeral capsule is a hallmark. Clinically, it presents as pain, stiffness, and dysfunction of the affected shoulder. Adhesive capsulitis is thought to afflict between 2 and 5% of the general population, with women affected more frequently than men. Individuals of middle age are most often affected, typically during the 5th to 7th decades of life.

Muscle energy techniques is a manual therapy that uses the gentle muscle contractions to relax and lengthen muscles and normalize joint motion. It is a class of soft tissue osteopathic manipulation consisting of isometric contraction designed to improve musculoskeletal function and reduce pain. The application of MET relaxes and improves biomechanics and result in improving functional ability.

Although conventional physical therapy treatment are used to treat frozen shoulder and effectiveness of muscle energy technique is proven, but the effect of first rib mobilization and MET has not been studied.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40-70 years
* Gender (both male and female)
* Subjects with adhesive capsulitis stage (II and III)

Exclusion Criteria:

* Previous surgery on affected shoulder
* Recent trauma to shoulder
* fracture

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale for pain | 3 weeks
  Scale consists of 4 questions regarding actual pain level, zero indicates no pain and 10 indicates worst pain imaginable
shoulder pain and disability index for shoulder pain | 3 weeks
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use.

SECONDARY OUTCOMES:
goniometer for measuring shoulder ranges | 3 weeks
  it is used to measure shoulder ranges such as flexion, abduction , internal and external rotation

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sanaullah, MS, Principal Investigator — Study Principal Investigator
Locations (1):
- Rabia welfare hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No